CLINICAL TRIAL: NCT03623698
Title: A Chart Review Assessing the Effects of Nebulised Hypertonic Saline on Respiratory-related Complications in Children and Young People With Neuromuscular Disease and Cerebral Palsy
Brief Title: Nebulised Hypertonic Saline in Children and Young People With Neuromuscular Disease and Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18IC4403
Record Dates: First submitted 2018-07-16; First posted 2018-08-09 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Neuromuscular Diseases
Keywords: Hypertonic saline; nebulised; children; young people; adolescents; respiratory
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before treatment: Children and young people with neuromuscular disease during the 12 months before being prescribed treatment with nebulised saline (0.9% - 7%)
- After treatment: Children and young people with neuromuscular disease during the 12 months after being prescribed treatment with nebulised saline (0.9% - 7%)
  Interventions: Drug: Nebulised hypertonic saline

INTERVENTIONS:
Drug: Nebulised hypertonic saline — Nebulised hypertonic saline used for a period of at least 12 months
  Other Names: 3% Sodium Chloride; 5% Sodium Chloride; 7% Sodium Chloride
  Groups: After treatment

SUMMARY:
Pneumonia, respiratory exacerbations, and chronic pulmonary infection are important causes of emergency admissions, hospitalisations and death in children with Neuromuscular disorders and Cerebral Palsy. Hence, there is a need for research on how to therapeutically aid airway clearance and decrease respiratory exacerbations. Studies have shown that nebulised Hypertonic Saline is well tolerated, reduces pulmonary exacerbations and improves lung function and Lung Clearance Index in patients with Cystic Fibrosis, and enhances mucociliary clearance in asthmatic patients. Nevertheless, to the investigators' knowledge, there is no available data concerning the use of nebulised Hypertonic Saline in the management of children with Neuromuscular disorders and Cerebral Palsy. This study aims to assess the effectiveness of nebulised Hypertonic Saline to decrease hospitalisations and courses of antibiotics in children with Neuromuscular disorders and Cerebral Palsy.

DETAILED DESCRIPTION:
Chart review of children and young people with Neuromuscular disease or Cerebral Palsy who are cared for in the Royal Brompton Hospital and that have been treated with nebulised hypertonic saline for at least 12 months.

To further complement data from hospital records, two questionnaires will be applied. Parents of children who meet criteria will be asked to complete the following questionnaires:

1. The National Health and Nutrition Examination Survey (NHANES) for Hospitalisation and access to are - HUQ.010; and
2. Questionnaire on Hypertonic Saline treatment.

Children from 10 - 18 years will be asked to complete the Questionnaire on Hypertonic Saline treatment.

AIMS

1. Explore whether treatment with nebulised Hypertonic Saline in children with Neuromuscular disease or Cerebral Palsy decreases respiratory-related complications.
2. Evaluate whether the treatment with nebulised hypertonic saline in children with neuromuscular disease or cerebral palsy improves the ease of airway clearance.
3. Explore how parents of children with Neuromuscular disease and children with Cerebral Palsy perceive the treatment with nebulised hypertonic saline compared with previous management.

Sample Size:

The investigators aim to recruit 40 participants for each group, including children and young people and their parents or legal guardians, as this is a pilot study.

STATISTICAL ANALYSIS PLAN

* Univariate X2 analysis for categorical variables to investigate Courses of antibiotic treatment.
* Univariate X2 analysis for categorical variables to investigate Number of hospitalisations.
* Student t testing will be used to analyse nocturnal oxygenation and ventilation outcomes comparing one year before and after starting treatment with Hypertonic Saline.
* Independent t testing and Mann-Whitney U test to analyse Rate of decline in pulmonary function.
* Cox proportional hazard model to test differences in primary endpoints for different baseline FVC.
* Univarate analysis to analyse Ease of airway clearance.
* Univariate analysis on perception of treatment.

Data and all appropriate documentation will be stored for a minimum of 10 years after the completion of the study, including the follow-up period.

ETHICS APPROVAL The Study Coordination Centre has obtained approval from the Yorkshire & The Humber - Leeds West Research Ethics Committee (REC) and Health Regulatory Authority (HRA). The study also received confirmation of capacity and capability from each participating NHS Trust before accepting participants into the study or any research activity was carried out. The study will be conducted in accordance with the recommendations for physicians involved in research on human subjects adopted by the 18th World Medical Assembly, Helsinki 1964 and later revisions.

CONSENT Consent to enter the study must be sought from each participant only after a full explanation has been given, an information leaflet offered and time allowed for consideration. Signed participant consent should be obtained. The right of the participant to refuse to participate without giving reasons must be respected. After the participant has entered the study the clinician remains free to give alternative treatment to that specified in the protocol at any stage if he/she feels it is in the participant's best interest, but the reasons for doing so should be recorded. In these cases the participants remain within the study for the purposes of follow-up and data analysis. All participants are free to withdraw at any time from the protocol treatment without giving reasons and without prejudicing further treatment.

CONFIDENTIALITY The Chief Investigator will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act.

PUBLICATION POLICY Data ownership rights will lie with the institution. Findings of this study will be presented as a Dissertation and will be available through Open Access. The investigators aim to publish findings in peer-review journals.

ELIGIBILITY:
Inclusion Criteria:

* Children with Neuromuscular disease or Cerebral Palsy who have been on treatment with nebulised Hypertonic Saline for at least 12 months.

Exclusion Criteria:

* Children also diagnosed with cystic fibrosis.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with Neuromuscular disease or Cerebral Palsy who have their care at the Royal Brompton Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Galaz Souza, Professional, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data ownership rights will lie with the institution.

REFERENCES:
- [Background] Allen J. Pulmonary complications of neuromuscular disease: a respiratory mechanics perspective. Paediatr Respir Rev. 2010 Mar;11(1):18-23. doi: 10.1016/j.prrv.2009.10.002. Epub 2009 Dec 2. PMID 20113987
- [Background] Lo Mauro A, Aliverti A. Physiology of respiratory disturbances in muscular dystrophies. Breathe (Sheff). 2016 Dec;12(4):318-327. doi: 10.1183/20734735.012716. PMID 28210319
- [Background] Boitano LJ. Management of airway clearance in neuromuscular disease. Respir Care. 2006 Aug;51(8):913-22; discussion 922-4. PMID 16867201
- [Background] Gerdung CA, Tsang A, Yasseen AS 3rd, Armstrong K, McMillan HJ, Kovesi T. Association Between Chronic Aspiration and Chronic Airway Infection with Pseudomonas aeruginosa and Other Gram-Negative Bacteria in Children with Cerebral Palsy. Lung. 2016 Apr;194(2):307-14. doi: 10.1007/s00408-016-9856-5. Epub 2016 Feb 16. PMID 26883134
- [Background] Phillips MF, Quinlivan RC, Edwards RH, Calverley PM. Changes in spirometry over time as a prognostic marker in patients with Duchenne muscular dystrophy. Am J Respir Crit Care Med. 2001 Dec 15;164(12):2191-4. doi: 10.1164/ajrccm.164.12.2103052. PMID 11751186
- [Background] Bell CF, Kurosky SK, Candrilli SD. Muscular dystrophy-related hospitalizations among male pediatric patients in the United States. Hosp Pract (1995). 2015;43(3):180-5. doi: 10.1080/21548331.2015.1033375. Epub 2015 Apr 1. PMID 25833749
- [Background] Yuan JX, McGowan M, Hadjikoumi I, Pant B. Do children with neurological disabilities use more inpatient resources: an observational study. Emerg Themes Epidemiol. 2017 Apr 27;14:5. doi: 10.1186/s12982-017-0059-1. eCollection 2017. PMID 28465710
- [Background] Elkins MR, Bye PT. Mechanisms and applications of hypertonic saline. J R Soc Med. 2011 Jul;104 Suppl 1(Suppl 1):S2-5. doi: 10.1258/jrsm.2011.s11101. No abstract available. PMID 21719889
- [Background] Elkins MR, Robinson M, Rose BR, Harbour C, Moriarty CP, Marks GB, Belousova EG, Xuan W, Bye PT; National Hypertonic Saline in Cystic Fibrosis (NHSCF) Study Group. A controlled trial of long-term inhaled hypertonic saline in patients with cystic fibrosis. N Engl J Med. 2006 Jan 19;354(3):229-40. doi: 10.1056/NEJMoa043900. PMID 16421364
- [Background] Amin R, Subbarao P, Jabar A, Balkovec S, Jensen R, Kerrigan S, Gustafsson P, Ratjen F. Hypertonic saline improves the LCI in paediatric patients with CF with normal lung function. Thorax. 2010 May;65(5):379-83. doi: 10.1136/thx.2009.125831. PMID 20435858
- [Derived] Galaz Souza N, Bush A, Tan HL. Exploratory study of the effectiveness of nebulised saline in children with neurodisability. Eur Respir J. 2021 Mar 18;57(3):2001407. doi: 10.1183/13993003.01407-2020. Print 2021 Mar. PMID 33184120

RESULTS

PARTICIPANT FLOW:
Groups:
- Children and Young People With Neuromuscular Disease: Children and young people with neuromuscular disease 18 years old or younger, who had been at least 12 months on prescribed nebulised saline (0.9%, 3%, 6%, and/or 7%) between 2011 and 2019.
Period: Overall Study
Arm/Group | Children and Young People With Neuromuscular Disease
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Children and Young People With Neuromuscular Disease: Children and young people with neuromuscular disease before nebulised saline was prescribed to them.
Arm/Group | Children and Young People With Neuromuscular Disease
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 24
Diagnosis [Count of Participants; unit: Participants]
  SMA | 14
  Chromosomal myopathy | 1
  Myotubular myopathy | 2
  Nemaline Rod myopathy | 1
  Congenital muscular dystrophy | 2
  LGMD | 1
  Joubert syndrome | 1
  Muscle eye brain disease | 1
  Rett syndrome | 1
Other characteristics [Count of Participants; unit: Participants]
  Non-ambulant | 21
  Tracheotomised | 3
  Gastrostomy feeding | 17
  Scoliosis | 13
Other treatments and medical procedures [Count of Participants; unit: Participants]
  Antibiotic prophylaxus | 12
  Dornase alpha | 5
  Home mechanical ventilation | 16
  Mechanically assisted cough | 14
Tonicity of nebulised prescribed [Count of Participants; unit: Participants]
  Hypertonic saline only (3%, 6%, 7%) | 9
  Isotonic saline only (0.9%) | 4
  Combination of hypertonic and isotonic saline | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Antibiotic Courses
Description: Treatments due to respiratory exacerbations
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Population: Two participants had incomplete data for this outcome, and/or their parents could not recall
Measure: Median (Inter-Quartile Range); unit: Courses of antibiotics
Groups:
- Before Treatment: Children and young people with neuromuscular disease during the 12 months before being prescribed treatment with nebulised saline
- After Treatment: Children and young people with neuromuscular disease during the 12 months after being prescribed treatment with nebulised saline (0.9%, 3%, 6%, and/or 7%)
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 22 | 22
Courses of antibiotics
  Total courses of antibiotics | 4 [2 to 6] | 1 [0 to 2]
  Courses of Oral antibiotics | 2.50 [1.00 to 6.00] | 1.00 [0.00 to 2.00]
  Courses of intravenous antibiotics | 1.00 [0.00 to 1.00] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: Before Treatment vs After Treatment; Statistical analysis was performed using IBM SPSS Statistics software, version 25. This analysis applies to the category of Total courses of antibiotics; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.500, 95% CI 2-sided [-4.000 to -1.500]
Statistical Analysis 2: Comparison: Before Treatment vs After Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Other — Linear mixed-effects model; p = 0.001, Mixed Models Analysis — 95% confidence interval, significance level p-values <0.05. Random effects pre-defined from theory and published data, and AIC was were used to define the best model. Outcome measures: Courses of antibiotics; Fixed effect: nebulised saline treatment; Random effects: age, gender, mechanical ventilation, tracheostomy, gastrostomy, non-ambulant; Restricted Maximum Likelihood (REML) = -2.88, 95% CI 2-sided [-4.46 to -1.29]

2. Primary Outcome: Number of Hospitalsations Due to Respiratory Exacerbations
Description: Number of respiratory exacerbations that required not planned hospitalisation
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Population: 23/24 patients were analysed for this outcome, because one patient had incomplete records on hospitalisations.
Measure: Median (Inter-Quartile Range); unit: Hospitalisations
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 23 | 23
Hospitalisations | 1 [0 to 2] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Before Treatment vs After Treatment; Statistical analysis was performed using IBM SPSS Statistics software, version 25; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.00, 95% CI 2-sided [-1.50 to -0.50]
Statistical Analysis 2: Comparison: Before Treatment vs After Treatment; Statistical analysis was performed using IBM SPSS Statistics software, version 25; Test type: Other; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]; Random effects: age, gender, prolonged mechanical ventilation (nasal or tracheostomy), and antibiotic prophylaxis; Restricted Maximum Likelihood (REML) = -1.02, 95% CI 2-sided [-1.53 to -0.52]

3. Secondary Outcome: Participant's Perception of Treatment
Description: Questionnaire: "Hypertonic saline treatment questionnaire". Perception of overall usefulness of nebulised hypertonic saline: "Useful", "Not useful", "I don't know".
Time Frame: At 12 months after starting treatment with hypertonic saline
Population: Applied to all participants aged 10-15 years who were able to communicate their views.
Measure: Count of Participants; unit: Participants
Arm/Group | Children and Young People With Neuromuscular Disease
Number analyzed (Participants) | 11
Participants
  Useful | 11
  Not useful | 0
  I don't know | 0

4. Secondary Outcome: Parent's or Legal Guardian's Perception of Treatment
Description: "Hypertonic saline treatment questionnaire for legal guardian". Measures the perception of overall usefulness of nebulised hypertonic saline through a likert scale: Very useful, useful, neither useful or not useful, not useful, not at all useful.
Time Frame: At 12 months after starting treatment with hypertonic saline
Measure: Count of Participants; unit: Participants
Groups:
- Parent's or Legal Guardians: One parent or legal guardian for each of the study participants
Arm/Group | Parent's or Legal Guardians
Number analyzed (Participants) | 24
Participants
  Very useful | 15
  useful | 9
  neither useful or not useful | 0
  not useful | 0
  not at all useful | 0

5. Secondary Outcome: Score on the Ease of Airway Clearance Pictorial Analogue Scale From Children and Young Adults as Participants
Description: Pictorial visual scale "Facial Rating of perceived exertion Scale". Measures ease of airway clearance. Values range starting in 0 (Extremely easy) to 10 (Extremely hard), including 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10. Numbers are also associated with facial expressions.
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 11 | 11
score on a scale | 6.45 [4 to 9] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Before Treatment vs After Treatment; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -4.50, 95% CI 2-sided [-5.50 to -3.00]

6. Secondary Outcome: Score on the Ease of Airway Clearance From Parents or Legal Guardians
Description: Measures ease of airway clearance through a 1-5 likert scale: 1) Very easy, 2) Easy, 3) Neither easy nor difficult, 4) Not easy, 5) Not at all easy.
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Before Treatment: Parents of children and young people with neuromuscular disease during the 12 months before being prescribed treatment with nebulised saline (0.9% - 7%)
- After Treatment: Parents pf children and young people with neuromuscular disease during the 12 months after being prescribed treatment with nebulised saline (0.9% - 7%)
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 24 | 24
score on a scale | 4.21 [3 to 5] | 2.13 [1 to 3]
Statistical Analysis 1: Comparison: Before Treatment vs After Treatment; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -2.00, 95% CI 2-sided [-2.5 to -2.0]

7. Secondary Outcome: Apnea Index (AI)
Description: The number of apneas recorded during the study per hour of sleep
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Population: 3/24 patients had records for this outcome
Measure: Mean (Standard Deviation); unit: Events per hour of sleep
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 3 | 3
Events per hour of sleep | 4.87 (1.02) | 0.40 (0.4)

8. Secondary Outcome: AHI
Description: Nocturnal Apnoea Hipopnea index: total number of apnea events plus hypopnea events divided by the total number of minutes of actual sleep time and then multiplied by 60.
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Measure: Mean (Standard Deviation); unit: Events per hour of sleep
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 3 | 4
Events per hour of sleep | 8.53 (1.70) | 1.38 (0.99)

9. Secondary Outcome: %SpO2
Description: Nocturnal oxygen saturation
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Population: 21/24 patients had complete records for this outcome
Measure: Mean (Standard Deviation); unit: percentage of SpO2
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 21 | 21
percentage of SpO2 | 96.55 (1.92) | 96.53 (1.83)
Statistical Analysis 1: Comparison: Before Treatment vs After Treatment; Test type: Other; p = 0.97, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.69 to 0.76]

10. Secondary Outcome: Nocturnal ODI
Description: Oxygen desaturation index: Number of desaturations per hour of sleep
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Population: 21/24 patients had complete records for this outcome
Measure: Mean (Standard Deviation); unit: Events per hour of sleep
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 21 | 21
Events per hour of sleep | 4.26 (3.42) | 3.32 (3.33)
Statistical Analysis 1: Comparison: Before Treatment vs After Treatment; Test type: Other; p = 0.09, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-3.26 to 0.34]

11. Secondary Outcome: TcPCO2
Description: Nocturnal Transcutaneous Carbon Dioxide in kPa
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Population: 21/24 patients had complete records for this outcome
Measure: Mean (Standard Deviation); unit: Kilopascal (kPa)
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 21 | 21
Kilopascal (kPa) | 5.77 (0.95) | 6.00 (1.04)
Statistical Analysis 1: Comparison: Before Treatment vs After Treatment; Test type: Other; p = 0.65, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.38 to 0.38]

12. Secondary Outcome: FEV1/FVC %Predicted Rate of Decline
Description: Rate of decline per year of Tiffenau index
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Population: 5/24 patients had complete records for this outcome
Measure: Median (Inter-Quartile Range); unit: percentage of predicted
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 5 | 5
percentage of predicted | 97.37 [84.50 to 110.50] | 98.89 [92.00 to 109.00]

13. Secondary Outcome: FEV1% Predicted Rate of Decline
Description: Rate of decline of Forced Expiratory Volume in first second (FEV1) percentage of predicted.
  Rate of decline is a measure of slope of FEV1 percentage predicted.
  Baseline slope: [(FEV1% at baseline / FEV1% 12 months before treatment) - 1] * 100 After treatment slope: [(FEV1% 12 months after treatment / FEV1% at baseline) - 1] * 100
Time Frame: Change from the baseline (before treatment) and 12 months after treatment
Measure: Median (Inter-Quartile Range); unit: percentage of predicted
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 2 | 5
percentage of predicted | -8.03 [-8.67 to -8.03] | 4.00 [-2.14 to 17.55]

14. Secondary Outcome: FVC% Predicted Rate of Decline
Description: Rate of decline of Forced Vital Capacity (FVC) percentage of predicted. Rate of decline is a measure of slope of FVC%.
  Baseline slope: [(FVC% at baseline / FVC% 12 months before treatment) - 1] * 100 After treatment slope: [(FVC% 12 months after treatment / FVC% at baseline) - 1] * 100
Time Frame: Change from baseline (before treatment) and 12 months after treatment
Measure: Median (Inter-Quartile Range); unit: percentage of predicted
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 2 | 3
percentage of predicted | -7.44 [-9.33 to -7.44] | 7.00 [-15.43 to 7.00]

15. Secondary Outcome: Peak Expiratory Flow (PEF)
Description: Peak expiratory flow percentage of predicted
Time Frame: Change from baseline peak expiratory flow at 12 months after starting treatment with hypertonic saline
Measure: Median (Inter-Quartile Range); unit: percentage of predicted
Arm/Group | Before Treatment | After Treatment
Number analyzed (Participants) | 6 | 5
percentage of predicted | 43.5 [33 to 47.5] | 47 [42 to 74]

ADVERSE EVENTS:
Time Frame: This was a retrospective study. Adverse events data was not collected.
Description: This was a retrospective study. Adverse events data was not collected.
Arm/Group | Children and Young People With Neuromuscular Disease
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This was a retrospective study, with potential for bias from self-selection. Each patient was used as their own control. The use of questionnaires had the potential for recall bias. This study did not have adherence data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT03623698/Prot_SAP_ICF_000.pdf